CLINICAL TRIAL: NCT00004584
Title: Safety and Antiviral Efficacy of a Novel HIV-1 Protease Inhibitor, BMS-232632, in Combination Regimen(s) as Compared to a Reference Combination Regimen(s) in Antiretroviral-Experienced HIV-Infected Subjects
Brief Title: Safety and Effectiveness of a New Protease Inhibitor, BMS-232632, in HIV-Positive Patients Who Have Received Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: 302B; AI424-009
Record Dates: First submitted 2000-02-10; First posted 2001-08-31 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Saquinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir; Saquinavir

INTERVENTIONS:
Drug: Atazanavir
Drug: Ritonavir
Drug: Saquinavir

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of an experimental protease inhibitor (a type of anti-HIV drug) called BMS-232632. Doctors will compare an anti-HIV drug combination that includes BMS-232632 to a drug combination that includes ritonavir.

DETAILED DESCRIPTION:
This is a three-arm study; patients are randomized to receive BMS-232632 at two different doses or RTV in combination with SQV and two nucleoside analogues over 48 weeks. Randomization is stratified for baseline phenotypic sensitivity.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load (level of HIV in the blood) of at least 2,000 copies/ml.
* Have a CD4 count of at least 100 cells/mm3 (or at least 75 cells/mm3 in patients who have never had an AIDS-defining illness).
* Are currently receiving an anti-HIV drug combination that includes a protease inhibitor or nonnucleoside reverse transcriptase inhibitor (NNRTI), and they have been taking this drug combination for at least 24 weeks. They must have responded well to this treatment at first (their viral load decreased) but are currently experiencing an increase in viral load.
* Will most likely respond well to the study drugs, as shown by the results of a lab test.
* Are at least 18 years old.
* Agree to use effective barrier methods of birth control (such as condoms).
* Are available for follow-up for at least 48 weeks.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a newly diagnosed opportunistic (HIV-related) infection requiring treatment.
* Have only recently become HIV positive.
* Abuse alcohol or drugs.
* Have severe diarrhea within 30 days of study entry.
* Have hemophilia.
* Have a history of pancreatitis.
* Have hepatitis within 30 days of study entry.
* Have peripheral neuropathy (a painful condition affecting the nervous system).
* Are unable to take medications by mouth.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (20):
  - Sorra Research Ctr / Med Forum, Birmingham, Alabama
  - AIDS Healthcare Foundation, Los Angeles, California
  - Robert Scott MD, Oakland, California
  - Univ of California - Davis Med Ctr / CARES, Sacramento, California
  - Avalar Medical Group, Tarzana, California
  - Yale Univ School of Medicine / AIDS Program, New Haven, Connecticut
  - Community Research Initiative of South Florida, Coral Gables, Florida
  - HIV Clinical Research, Fort Lauderdale, Florida
  - Infectious Disease Research Institute, Tampa, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Louisiana State Univ Med Ctr / HIV Outpatient Clinic, New Orleans, Louisiana
  - Albany Med College, Albany, New York
  - St Vincents Hosp / Clinical Research Program, New York, New York
  - Univ Hosps of Cleveland, Cleveland, Ohio
  - The Research and Education Group, Portland, Oregon
  - Julio Arroyo, West Columbia, South Carolina
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Texas Tech Health Sciences Ctr, El Paso, Texas
  - Houston Clinical Research Network / Div of Montrose Clinic, Houston, Texas
- Canada (3):
  - Ottawa General Hospital, Ottawa, Ontario
  - Toronto Hosp, Toronto, Ontario
  - Montreal Chest Institute, Montreal, Quebec
- France (7):
  - Hopital Pellegrin Tripode, Bordeaux
  - Hopital De L'Hotel Dieu, Nantes
  - Hopital De L'Archet 1, Nice
  - Srev Du Pr Gentilini, Paris
  - Hopital De Haut Leveque, Pessac
  - Hospital Gustave Dron, Tourcoing
  - Hopital Paul Brousse, Villejuif
- Germany (3):
  - Brennerstr 71, Hamburg
  - Georg-Str 46, Hanover
  - Praxisgemeinschaft, Munich
- Italy (5):
  - Reparto Malattie Infettive, Antella
  - Clinical Malattie Infettive, Milan
  - Ospedale Luigi Cacco Moroni, Milan
  - Clinical Malattie Infettive / Univ Modena, Modena
  - Ospedale degli Infermi, Rimini

REFERENCES:
- [Background] Haas DW, Zala C, Schrader S,Thiry A, McGovern R, Schnittman S. AI424009: Atazanavir plus Saquinavir once daily favorably affects total cholesterol (TC), fasting triglyceride (TG), and fasting LDL cholesterol (LDL) profiles in patients failing prior therapy week 48. 9th Conf on Retroviruses and Opportunistic Infect. 2002 Feb 24-28 (abstract no 42)
- [Background] Haas DW, Zala C, Schrader S,Thiry A, McGovern R, Schnittman S. AI424-009: Once-Daily Atazanavir plus Saquinavir favorably affects total cholesterol and fasting triglycerides in patients failing prior PI therapy study BMS-009,week 24. 41st Annual Conf on Antimicrobial Agents and Chemotherapy. 2001 Feb 16-19 (abstract no LB-16)